CLINICAL TRIAL: NCT04300790
Title: Study to Evaluate the Effect of Metformin in the Prevention of Hyperglycemia in HR[+]/HER2[-] PIK3CA-mutation Advanced Breast Cancer Patients Treated With Alpelisib Plus Endocrine Therapy. Study Metallica
Brief Title: Study to Evaluate the Effect of Metformin in the Prevention of HG in HR[+]/HER2[-] PIK3CA-mut Advanced BC Patients
Acronym: METALLICA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedSIR (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEDOPP240; 2019-003970-26 (EudraCT Number)
Record Dates: First submitted 2020-02-11; First posted 2020-03-09 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer
Keywords: ER; PI3KMut; HER2; Metastatic; unresectable; breast; hyperglycemia; men
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis; Hyperglycemia; Multiple Endocrine Neoplasia Type 1 | interventions — Alpelisib; Metformin; Fulvestrant; Letrozole; exemestane; Vildagliptin; Tamoxifen

STUDY DESIGN:
Intervention Model Description: This is a multicenter, open-label, three-cohort, Simon's two stage design, phase II clinical trial.
  Cohort A: Normal fasting glycemia < 100 mg/dL and HbA1c < 5,7: 48 patients (20 stage 1 + 28 stage 2). Patients in cohort A will receive.
  Cohort B: fasting glycemia 100 mg/dL (5.6 mmol/L) to 140mg/dL (7.8 mmol/L). 20 patients (7 stage 1 + 13 stage 2).
  Cohort C: T2DM diagnosed clinically ≥ 90 days prior to screening, HbA1c < 7,5 %, insulin naïve (5 during stage I + 15 during stage II).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CohortA: Normoglycemic patients (Experimental): Alpelisib plus metformin and Endocrine Therapy (fulvestrant or Letrozole or Exemestane): During the first cycle, patients will receive Endocrine Therapy and metformin at least one-week prior alpelisib administration (D8).
  Alpelisib (BYL719) 300 mg PO (two tablets of 150 mg once a day) on a continuous dosing schedule starting on Cycle 1.
  Metformin 500 mg BID with breakfast and dinner. After 3 days, if no GI intolerance, increase to 1000 mg BID with breakfast and dinner. If not tolerated, reduce to prior tolerated dose. Titrate to 1000mg BID over a period of at least 4 additional days.
  Endocrine Therapy:
  Fulvestrant 500 mg (intramuscular injection) on days 1 and 15 of cycle 1 (28 days); then every 4 weeks as per SoC- (day 1 of subsequent 28-days cycles) or Letrozole 2,5 mg, once daily, orally or Exemestane 25 mg once daily, orally.
  Interventions: Drug: Alpelisib; Drug: Metformin; Drug: Fulvestrant; Drug: Letrozole; Drug: Exemestane
- CohortB: Pre-diabetic patients (Experimental): Alpelisib plus metformin and Endocrine Therapy (fulvestrant or Letrozole or Exemestane): During the first cycle, patients will receive Endocrine Therapy and metformin at least one-week prior alpelisib administration (D8). Alpelisib (BYL719) 300 mg PO (two tablets of 150 mg once a day) on a continuous dosing schedule starting on Cycle 1.
  Metformin 500 mg BID with breakfast and dinner. After 3 days, if no GI intolerance, increase to 1000 mg BID with breakfast and dinner. If not tolerated, reduce to prior tolerated dose. Titrate to 1000mg BID over a period of at least 4 additional days.
  Endocrine Therapy:
  Fulvestrant 500 mg (intramuscular injection) on days 1 and 15 of cycle 1 (28 days); then every 4 weeks as per SoC- (day 1 of subsequent 28-days cycles) or Letrozole 2,5 mg, once daily, orally or Exemestane 25 mg once daily, orally.
  Interventions: Drug: Alpelisib; Drug: Metformin; Drug: Fulvestrant; Drug: Letrozole; Drug: Exemestane
- CohortC: Insulin naïve type 2 diabetic mellitus patients (Experimental): Alpelisib plus metformin plus vildagliptin and Endocrine Therapy (fulvestrant or Letrozole or Exemestane or Tamoxifen): During the first cycle, patients will receive Endocrine Therapy, metformin and vildagliptin at least two-weeks prior alpelisib administration (D15).Alpelisib (BYL719) 300 mg PO (two tablets of 150 mg once a day) on a continuous dosing schedule starting on Cycle 1.
  Metformin 500 mg BID with breakfast and dinner. After 3 days, if no GI intolerance, increase to 1000 mg BID with breakfast and dinner. If not tolerated, reduce to prior tolerated dose. Titrate to 1000mg BID over a period of at least 4 additional days.
  Endocrine Therapy:
  Fulvestrant 500 mg (intramuscular injection) on days 1 and 15 of cycle 1 (28 days); then every 4 weeks as per SoC- (day 1 of subsequent 28-days cycles) or Letrozole 2,5 mg, once daily, orally or Exemestane 25 mg once daily, orally or Tamoxifen 20 mg once daily, orally.
  Interventions: Drug: Alpelisib; Drug: Metformin; Drug: Fulvestrant; Drug: Letrozole; Drug: Exemestane; Drug: Vildagliptin; Drug: Tamoxifen

INTERVENTIONS:
Drug: Alpelisib — Alpelisib (BYL719): starting dose at 300 mg/QD.; 2 tablets once a day, oral administration, continuously during 28-day cycles until disease progression or unacceptable toxicity.
  Other Names: BYL719
Drug: Metformin — 500 mg BID with breakfast and dinner. After 3 days, if no (GI) intolerance, increase to 1000 mg BID with breakfast and dinner. If not tolerated, reduce to prior tolerated dose. Titrate to 1000mg BID over a period of at least 4 additional days
Drug: Fulvestrant — fulvestrant (500 mg IM injections; loading dose 500mg every two weeks for the first month; then every 4 weeks as per standard of care [SoC].
  Patients should be started on metformin and fulvestrant within 7 to 14 days prior to start on alpelisib (D1C1)
Drug: Letrozole — Letrozole 2.5 mg tablets, once daily, orally
Drug: Exemestane — Exemestane 25 mg tablets, once daily, orally
Drug: Vildagliptin — Vildagliptin 50 mg tablets, twice daily, orally with breakfast and dinner
  Arms: CohortC: Insulin naïve type 2 diabetic mellitus patients
Drug: Tamoxifen — Tamoxifen 20 mg tablets, once daily, orally
  Arms: CohortC: Insulin naïve type 2 diabetic mellitus patients

SUMMARY:
Men and post- or induced menopausal women with ER[+] and/or PgR[+], HER2[- ] advanced BC, with centrally-confirmed PI3KCAMut who progressed to an aromatase inhibitor (AI) regimen.

DETAILED DESCRIPTION:
Men and post- or induced menopausal women with ER[+] and/or PgR[+], HER2[- ] advanced BC, with centrally-confirmed PI3KCAMut who progressed to an aromatase inhibitor (AI) regimen.Men and post- or induced menopausal women with ER[+] and/or PgR[+], HER2[- ] advanced BC, with centrally-confirmed PI3KCAMut who progressed to an aromatase inhibitor (AI) regimen.Measurable or evaluable disease according to RECIST v.1.1 criteria.No prior treatment with fulvestrant or PI3K, AKT or mTOR inhibitors.

No more than one prior line of chemotherapy for metastatic breast cancer (MBC). Eastern Cooperative Oncology Group (ECOG) Performance Status 0 - 1. Non-diabetic patients will be assigned to Cohorts A or B and insulin naïve patients with established diagnosis of type 2 diabetes mellitus will be assigned to Cohort C.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form (ICF)prior to participation in any study- related activities.
2. Men, pre-menopausal or post-menopausal women ≥ 18 years of age at the time of signing ICF.
3. Men and pre-menopausal women should have been treated with a luteinizing hormone-releasing hormone (LHRH) analogue at least one week prior to study entry. Post-menopausal women are defined as per the following criteria:

   * Age 3 60 years, or
   * Age < 60 years and cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; and serum estradiol and/or follicle stimulating hormone (FSH) level within the laboratory's reference range for postmenopausal females; or documented bilateral oophorectomy.
4. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
5. Histologically proven diagnosis of advanced breast cancer (ABC, loco regionally recurrent not amenable to curative therapy or metastatic disease).
6. Confirmed diagnosis of estrogen receptor (ER)[+] and/or progesterone receptor (PR)[+] (with ≥1% positive stained cells according to National Comprehensive Cancer Network [NCCN] and American Society of Clinical Oncology [ASCO] guidelines) and human epidermal growth factor receptor 2 (HER2)-negative (0 or 1+ by immunohistochemistry [IHC] or 2+ and negative by in situ hybridization [ISH] test) breast cancer in the advanced setting.
7. Measurable or evaluable disease as per Response Evaluation Criteria in Solid Tumors (RECIST) version (v.)1.1 criteria. Patients with bone- only metastases are eligible.

   Patients with no measurable or evaluable disease will be considered by the study medical monitor.
8. Presence of phosphatidylinositol-4,5-bisphosphate 3-kinase catalytic subunit alpha (PIK3CA)-mutated (PIK3CAMut) determined on the most recent tumor tissue specimen (frozen or formalin-fixed paraffin- embedded [FFPE]) or plasma circulating tumor DNA (ctDNA).

   Note: Prior tests of PIK3CAMut preceding the ICF signature will be considered valid if the results are documented and captured in the medical record during the pre-screening period. If the PIK3CA status is unknown, tumor tissue can be provided during pre-screening phase to assess the presence of PIK3CAMut. In case when tumor tissue specimen cannot be obtained, presence of PIK3CAMut can be carried out on plasma in the pre-screening period prior to initiate the study treatment.
9. No more than 2 prior lines of endocrine therapy for ABC. Regimen with documented evidence of progression while on (neo)adjuvant endocrine therapy or within the first 12 months from completion of (neo)adjuvant endocrine therapy will be considered as a prior line.
10. Patients who progressed with documented evidence of progression while on or after an aromatase inhibitors (AI)-based regimen for metastatic disease, or who relapsed with documented evidence of progression while on (neo)adjuvant AI-based regimen or within the first 12 months from completion of (neo)adjuvant AI-based regimen.
11. PPatients are permitted to have received previous fulvestrant either as (neo)adjuvant regimen or as first-line regimen for metastatic disease.

    Note 01: Patients with secondary resistance (relapse while on adjuvant endocrine therapy but after the first 2 years, or relapse within 12 months of completing adjuvant endocrine therapy, or progression ≥ 6 months after initiating endocrine therapy for metastatic disease, while on endocrine therapy) to fulvestrant will be treated with either fulvestrant, letrozole, exemestane or tamoxifen based on physician's criteria. Patients with primary endocrine resistance (relapse while on the first 2 years of adjuvant endocrine therapy, or progression within first 6 months of first-line endocrine therapy for metastatic disease, while on endocrine therapy) to fulvestrant would be treated with either letrozole or exemestane based on physician's criteria.

    Note 02: Anti-estrogens in current development (i.e. SERMs, SERDs, PROTAC, etc.) are allowed to be used as (neo)adjuvant regimen or as first-line regimen for metastatic disease according to investigator criteria.
12. Received no more than 1 prior regimen of chemotherapy in the metastatic setting. Regimen with documented evidence of progression while on (neo)adjuvant chemotherapy or within the first 6 months from completion will be considered as a prior line.
13. For Cohort A and B only; Fasting plasma glucose (FPG) and glycosylated hemoglobin (HbA1c):

    Cohort A: FPG ≤100 mg/dL (5.6 mmol/L) and HbA1c < 5,7

    Cohort B: FPG 100-140 mg/dL (5,6-7,8 mmol/L) (impaired fasting glucose values) or HbA1c 5,7-6,4%.
14. For Cohort C only:

    * T2DM subjects diagnosed clinically ≥ 90 days prior to screening,
    * HbA1c < 7,5%.
    * Stable diabetes treatment for 90 days prior to screening
15. If central nervous system (CNS) metastases are present, controlled local disease without corticoids and/or anti-epileptic medication is required.
16. Adequate bone marrow and organ function as defined by the following laboratory values:

    * Hematological:

      * White blood cell (WBC) count ≥ 3.0 x 109/L; absolute neutrophil count (ANC) > 1.5 x 109/L; platelet count > 100.0 x109/L; and hemoglobin > 9.0 g/dL.
      * Calcium(correctedforserumalbumin)andmagnesiumwithin normal limits or ≤ grade 1 according to National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) v.4.03 if judged clinically not significant by the investigator. Potassium within normal limits or corrected with supplements.
      * International normalized ratio (INR) ≤1.5.
    * Hepatic:

      * Bilirubin < 2 times the upper limit of normal (× ULN). Any elevated bilirubin should be asymptomatic at enrollment except for patients with Gilbert's disease who may be only included if the total bilirubin is ≤ 3 x ULN or direct bilirubin ≤ 1.5 x ULN.
      * Aspartate transaminase (AST), and alanine transaminase (ALT) ≤ 3 times × ULN (in the case of liver metastases ≤ 5 × ULN, stable for 2 weeks, without the evidence of biliary obstruction by imaging).
    * Renal:

      * Creatinine clearance ≥ 35 mL/min using Cockcroft-Gault formula.

    Other:
    * Fasting serum amylase ≤ 2 × ULN and fasting serum lipase below or equal to ULN.
    * FPG ≤ 140 mg/dL (7,7 mmol/L) and HbA1c ≤ 6,4% (both criteria must be met for Cohorts A and B only).
17. Patients who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
18. Resolution of all acute toxic effects of prior anti-cancer therapy to grade £ 1 as determined by the NCI-CTCAE v.4.03 (except for alopecia or other toxicities, such as myelosuppression, not considered a safety risk for the patient at investigator's discretion).

Exclusion Criteria:

1. Prior treatment with a phosphatidylinositol 3-kinase (PI3K), AKT, or mammalian target of the rapamycin (mTOR) inhibitor. Prior treatment with a cyclin-dependent kinase 4/6 inhibitor (CDK4/6i) is allowed.
2. Known hypersensitivity to alpelisib, fulvestrant, letrozole, exemestane, tamoxifen or to any of their excipients.
3. Patients treated with insulin.
4. Cohort A and B; Established diagnosis of type 1 or 2 diabetes mellitus (DM) requiring anti-diabetic drugs. Patients with an impaired FPG or HbA1c as per inclusion criterion #14 are eligible to enter the cohort B if no anti-diabetic drug were received in the last 14 days prior to the start of study treatment.
5. Cohort C;

   * Type 1 diabetes patients.
   * Renal impairment defined as eGFR < 25 mL/min/1.73 m2 as per CKD-EPI.
   * History of proliferative retinopathy or maculopathy requiring acute treatment.
   * History of pancreatitis (acute or chronic).
   * Severe neuropathy, in particular autonomic neuropathy, i.e. gastroparesis, as judged by the investigator.
   * History of ketoacidosis or hyperosmolar state episodes.
   * History of intolerance to antidiabetic drugs except metformin.
6. Inflammatory breast cancer at screening.
7. Concurrent malignancy or malignancy within first 3 years of start of study treatment, except for adequately treated, basal or squamous cell carcinoma, non-melanomatous skin cancer, or curatively resected cervical cancer.
8. Past medical history of acute or chronic pancreatitis within one year prior to screening.
9. Impaired gastrointestinal (GI) function or GI disease that may affect the absorption of study drugs (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection) based on investigator's discretion.
10. Documented pneumonitis/interstitial lung disease (the chest computed tomography [CT] scan performed at baseline for the purpose of tumor assessment should be reviewed to confirm that there are no relevant pulmonary complications present.
11. Patients with Child-Pugh score B or C liver disease.
12. Patients with renal failure
13. Patients with unresolved osteonecrosis of the jaw.
14. History of Stevens-Johnson Syndrome (SJS), erythema multiforme (EM), toxic epidermal necrolysis (TEN) or Drug Reaction with Eosinophilia and Systemic Symptoms (DRESS).
15. Uncontrolled hypertension defined by a Systolic Blood Pressure (SBP) ≥ 160 mm Hg and/or Diastolic Blood Pressure (DBP) ≥ 100 mm Hg, with or without anti-hypertensive medication. Initiation or adjustment of antihypertensive medication(s) is allowed prior to screening.
16. Clinically significant uncontrolled heart disease and/or recent cardiac events including any of the following:

    1. History of angina pectoris, coronary artery bypass graft (CABG), symptomatic pericarditis, or myocardial infarction within 6 months prior to the start of study treatment.
    2. History of documented congestive heart failure (New York Heart Association functional classification III-IV).
    3. Left Ventricular Ejection Fraction (LVEF) < 50% at screening as determined by Multiple Gated acquisition (MUGA) scan or echocardiogram (ECHO).
    4. Clinically significant cardiac arrhythmias, (e.g., ventricular tachycardia), complete left bundle branch block, high grade AV block (e.g., bifascicular block, Mobitz type II, and third-degree AV block without pacemaker in place).
    5. Long QT syndrome, family history of idiopathic sudden death or congenital long QT syndrome, or Fredericia QT correction formula (QTcF) > 470msec at screening (mean of triplicate ECGs).
17. Any other concurrent severe and/or uncontrolled medical condition that would, in the investigator's judgment, contraindicate subject participation in the clinical study (e.g., chronic active hepatitis [testing not mandatory unless required by local regulations or requirements], severe hepatic impairment, etc.).
18. Treatment with any of the following medications and cannot be discontinued seven days prior to the start of the treatment:

    * Strong inhibitors or inducers of the isoenzyme cytochrome P450 3A (CYP3A) within the last 5 days prior to study entry.
    * Inhibitors of breast cancer resistance protein (BCRP).
19. Radiotherapy ≤ four weeks or limited field radiation for palliation ≤ two weeks prior to study treatment start, and who has not recovered to grade 1 or better from related side effects of such therapy (except for alopecia).
20. Patient is currently receiving or has received systemic corticosteroids ≤ 2 weeks prior to study treatment start or who have not fully recovered from side effects of such treatment.

    Note: The following uses of corticosteroids are permitted: single doses, topical applications (e.g., for rash), inhaled sprays (e.g., for obstructive airways diseases), eye drops or local injections (e.g., intra-articular).
21. Participation in a prior investigational study within 30 days prior to the start of study treatment or within five half-lives of the investigational product, whichever is longer.
22. Patient has not recovered from all toxicities related to prior anticancer therapies to NCI-CTCAE version 4.03 grade ≤1. Exception to this criterion: subjects with any grade of alopecia are allowed to enter the study.
23. Known history of Human Immunodeficiency Virus (HIV) infection.
24. Any other concurrent severe and/or uncontrolled medical condition that would, in the investigator's judgment, contraindicate subject participation in the clinical study (e.g., chronic active hepatitis, severe hepatic impairment).
25. Patient is a breastfeeding or pregnant woman as confirmed by a positive serum (hCG) or urine test prior to initiating study treatment.
26. Women of child-bearing potential defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during study treatment and for at least 1 year after stopping fulvestrant or for at least 1 week after stopping alpelisib. Highly effective contraception methods include:

    * Total abstinence (when this is in line with the preferred and usual lifestyle of the subject). Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy or bilateral tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
    * Male sterilization (at least six months prior to screening). For female subjects on the study the vasectomized male partner should be the sole partner for that subject.
    * Combination of the following:
    * Placement of intrauterine device (IUD) or intrauterine system (IUS)
    * Use of diaphragm or cervical caps by the patient herself or condom by the male partner combined with use of spermicidal products/vaginal suppository. Note: Use of hormonal methods of contraception (estrogen and progesterone) or hormonal replacement therapy are not allowed in the study.

    Note: Women are considered postmenopausal and not of childbearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (i.e., age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy, or bilateral tubal ligation at least 6 weeks before taking study treatment. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is, she considered not of childbearing potential.
27. Patient is a sexually active male not sterilized (at least 6 months prior to screening) or unwilling to use a condom during intercourse while taking study treatment, and for at least 1 year after stopping fulvestrant or for at least 1 week after stopping alpelisib. A condom is required for all sexually active male participants to prevent them from fathering a child AND to prevent delivery of study treatment via seminal fluid to their partner. In addition, male participants must not donate sperm during study and up to the period specified above.

Note: If local regulations to prevent pregnancy deviate from the contraception methods listed above, local regulations apply and will be described in the ICF.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2020-10-23 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2025-03-16 (Actual)

PRIMARY OUTCOMES:
Assess the rate of patients with G3-4 hyperglycemia (HG) by CTCAE v4.03 over the first 2 cycles of treatment with alpelisib (BYL719) (Cohorts A and B) | Baseline up tp 15 months
  The primary objective is to assess the rate of patients with G3-4 (CTCAE v4.03) hyperglycemia (HG) over the first 2 cycles of treatment with alpelisib (BYL719) (300 mg/QD) plus endocrine therapy and metformin, in patients with normal fasting glycemia and HbA1c (cohort A), and in patients with high-risk criteria (cohort B).
Assess the rate of patients with permanent discontinuation of alpelisib due to related AEs after 8 weeks of treatment with alpelisib plus endocrine therapy and antidiabetic treatment (Cohort C). | Baseline up tp 15 months
  The primary objective is to assess the rate of patients with permanent discontinuation of alpelisib due to related AEs after 8 weeks of treatment with alpelisib plus endocrine therapy and antidiabetic treatment in patients with insuline naive type 2 diabetic mellitus patients (cohort C).

SECONDARY OUTCOMES:
Clinical efficacy of alpelisib plus endocrine therapy, and antidiabetic treatment will be exploratory evaluated based on CTCAE V4.03 guidelines | Baseline up to 15 months
  To evaluate the clinical efficacy -in terms of progression-free survival (PFS), overall response rate (ORR), time to response (TTR), duration of the response (DoR), time to progression (TTP), clinical benefit rate (CBR)- of combining alpelisib plus endocrine therapy, and antidiabetic treatment in patients with HR[+]/HER2[-], PIK3CAMut ABC in all study cohorts and according to the different endocrine agent received.
Progression free survival [PFS] | Baseline up to 15 months
  Progression free survival [PFS] (defined as the time from the date of inclusion to the date of the first documented progression or death due to any cause, in the overall population, in all cohorts, and according to the different endocrine agent received. If a patient has not had an event, PFS will be censored at the date of the last adequate tumor evaluation [see RECIST 1.1]).
Overall response rate [ORR] | Baseline up to 15 months
  Overall response rate [ORR] (defined as the proportion of patients with best overall response -including complete response [CR] or partial response [PR]- based on local investigator's assessment (RECIST 1.1), in the overall population, in all cohorts, and according to the different endocrine agent received.
Time to response [TTR] | Baseline up to 15 months
  Time to response [TTR], defined as the period from the treatment initiation to time of the first objective tumor response (tumor shrinkage of ≥ 30%) observed for patients who achieved a CR or PR, as determined locally by the investigator through the use of RECIST v.1.1.· in all the cohorts, and according to the different endocrine agent received).
Duration of the response [DoR] | Baseline up to 15 months
  The period from the first occurrence of a documented objective response to disease progression or death from any cause, whichever occurs first, as determined locally by the investigator through use of RECIST v.1.1. in all the cohorts, and according to the different endocrine agent received.
Time to progression [TTP] | Baseline up to 15 months
  Time to progression [TTP] (defined as the time from date of randomization/start of treatment to the date of event defined as the first documented progression or death due to underlying cancer, in the overall population, in all cohorts, and according to the different endocrine agent received. If a patient has not had an event, time to progression is censored at the date of last adequate tumor assessment).
Clinical benefit rate [CBR] | Baseline up to 15 months
  Clinical benefit rate [CBR] (defined as the proportion of patients with a best overall response of CR or PR or SD or Non-CR/Non-PD lasting more than 24 weeks based on local investigator assessment), in the overall population, in all cohorts, and according to the different endocrine agent received.
Rate of any grade and grade 3-4 HG by CTCAE v.4.03 in Cohorts A, B, and C | Baseline up to 15 months
  To assess the rate of any grade and grade 3-4 HG by CTCAE v.4.03 in cohorts A, B, and C for Metallica and its comparation with Solar-1, and Bylieve trials.
Rate of patients with permanent treatment discontinuation at 8 weeks | Baseline up to 15 months
  To assess the rate of patients with permanent treatment discontinuation at 8 weeks of treatment with alpelisib due to treatment-related AEs in patients with normal fasting glycemia and HbA1c (Cohort A), and in patients with impaired fasting glucose criteria (Cohort B).
Rate of patients with permanent treatment discontinuation in all cohorts | Baseline up to 15 months
  To assess the rate of patients with permanent discontinuation due to alpelisib treatment-related AEs in Cohorts A, B, and C for Metallica, and to compare it with SOLAR-1, and Bylieve trials.
Rate of patients with permanent treatment discontinuation antidiabetic treatment), due to related AEs in all patients and all study cohorts | Baseline up to 15 months
  To assess the rate of patients with alpelisib permanent discontinuation due to related AEs over the first 8 weeks in the overall population, in all and according to the different endocrine agent received.
Rate of patients with grade 3-4 HG as per CTCAE v.4.03 over the first 8 weeks of treatment with alpelisib plus endocrine therapy and antidiabetic treatment and during the whole study | Baseline up to 15 months
  To assess the rate of patients with grade 3-4 HG as per CTCAE v.4.03 over the first 8 weeks of treatment with alpelisib plus endocrine therapy and antidiabetic treatment and during the whole study, in all study cohorts, according to the different endocrine agent received.
Rate of patients that requires insulin to control HG during the first 8 weeks and throughout study | Baseline up to 15 months
  To assess the rate of patients that requires insulin to control HG during over the first 8 weeks of treatment with alpelisib plus endocrine therapy and antidiabetic treatment and during the whole study, in all study cohorts, according to the different endocrine agent received.
  The number and class of antidiabetic agents used during the first 8 weeks and throughout study, in the overall population, in all the cohorts.
Type of HG in patients with grade 3-4 HG as per CTCAE v.4.03 and 5.0 | Baseline up to 15 months
  To define the type of HG in patients with grade 3-4 HG as per CTCAE v.4.03 and 5.0 in all the study cohorts and according to the different endocrine agent received, and the rate of patients with HG all the cohorts and according to the different endocrine agent received as per CTCAE v.4.03 and as per CTCAE v.5.
The rate of any grade and grade 3-4 diarrhea by CTCAE v.4.03 | Baseline up to 15 months
  To assess the rate of any grade and grade 3-4 diarrhea by CTCAE v.4.03 for Metallica.
Safety and tolerability of the combination of alpelisib with endocrine therapy, and antidiabetic treatment | Baseline up to 15 months
  To evaluate the safety and tolerability of the combination of alpelisib with endocrine therapy, and antidiabetic treatment in all study cohorts and according to the different endocrine agent received.
AEs according to the different endocrine agent received as per CTCAE v.4.03 | Baseline up to 15 months
  To define the rate of patients with grade 3-4 AEs as per CTCAE v.4.03 in all study cohorts and according to the different endocrine agent received.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Llombart, Principal Investigator — MedSIR
Locations (19):
- Spain (19):
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitari Vall D'Hebron, Barcelona
  - Institut Català d' Oncologia L'Hospitalet (ICO), Barcelona
  - Hospital Universitario de Basurto, Bilbao
  - Hospital Provincial de Castellón, Castellon
  - Hospital San Pedro de Alcántara, Cáceres
  - Onkologikoa, Donostia / San Sebastian
  - Hospital Universitario Clínico San Cecilio de Granada, Granada
  - Hospital Universitario Insular de Gran Canaria, Las Palmas de Gran Canaria
  - Hospital Universitario de Leon, León
  - Hospital Beata María Ana, Madrid
  - Hospital Ruber Internacional, Madrid
  - Hospital Universitario Doce de Octubre, Madrid
  - Hospital Universitario Sanchinarro, Madrid
  - Hospital Clínico Universitario Virgen de la Arrixaca, Murcia
  - Complejo Hospitalario Universitario de Santiago (CHUS), Santiago de Compostela
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
  - Instituto Valenciano de Oncología (IVO), Valencia

IPD SHARING:
Plan to Share IPD: No